CLINICAL TRIAL: NCT01936779
Title: Investigating Intra-hepatic Fatty Acid Partitioning and Its Regulation in Man. Studies to Understand the Role of Dietary Nutrients in Liver Fat Metabolism in Relation to Obesity in Man.
Brief Title: Understanding the Role of Dietary Fatty Acids on Liver Fat Metabolism in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Oxlip-2013
Record Dates: First submitted 2013-09-02; First posted 2013-09-06 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: NAFLD
Keywords: plasma triglycerides; dietary fat; liver fat metabolism; human
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary supplement: fatty acid active (Active Comparator): 4g/day n-3 fatty acids for 8 weeks
  Interventions: Dietary Supplement: Dietary supplement: fatty acid
- Dietary supplement: fatty acid placebo (Placebo Comparator): 4g/day olive oil for 8 weeks
  Interventions: Dietary Supplement: Dietary supplement: fatty acid

INTERVENTIONS:
Dietary Supplement: Dietary supplement: fatty acid — Consumption of n-3 fatty acids for 8 weeks
  Other Names: n-3 fatty acids (EPA and DHA)
  Arms: Dietary supplement: fatty acid active
Dietary Supplement: Dietary supplement: fatty acid — Consumption of olive oil for 8 weeks.
  Other Names: Olive oil
  Arms: Dietary supplement: fatty acid placebo

SUMMARY:
High levels of fatty substances in the blood increase the risk of developing heart disease. Investigators know a lot about one of these fatty substances, cholesterol. However, there is another fatty substance in the blood called triglyceride. Investigators do not understand much about what regulates the rate at which the liver produces triglyceride and liberates it into the bloodstream after eating a meal(s). It is known that taking fish oil lowers the amount of blood triglyceride however, it remains unclear how this happens. Investigators will study if changes in liver fat metabolism, after taking fatty acids found in fish oil (n-3 fatty acids)can explain the lowering of blood triglyceride. Investigators also want to know if taking fish oil alters the amount of fat that accumulates within the liver.

DETAILED DESCRIPTION:
Investigators will recruit men and women with no medical condition or relevant drug therapy that affects liver fat metabolism.

Purpose and design:

Investigators are asking the research question: "How do specific fatty acids, such as those found in fish ((n-3) fatty acids) influence postprandial liver fat metabolism?"

It is known that n-3 fatty acids lower plasma triglyceride concentrations but it remains unclear how this happens.

To address this research question investigators want to undertake detail physiological studies, in a randomised study where individuals will be studied before and after taking n-3 fatty acids or a placebo oil.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* BMI >19 <35kg/m2
* No medical condition or relevant drug therapy known to affect liver metabolism

Exclusion Criteria:

* Age <18 or >65 years
* Body mass index <19 or >35kg/m2
* A blood haemoglobin <120mg/dL
* Any metabolic condition or relevant drug therapy
* People allergic to fish / seafood or nuts
* Smoking
* History of alcoholism or a greater than recommended alcohol intake
* Pregnant or nursing mothers
* Women prescribed any contraceptive agent or device including oral contraceptives, hormone replacement therapy (HRT) or who have used these within the last 12 months
* History of severe claustrophobia
* Presence of metallic implants, pacemaker
* Haemorrhagic disorders
* Anticoagulant treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Plasma triglyceride concentrations | Eight weeks
  Investigators will measure plasma triglyceride concentrations at baseline and 8 weeks after taking n-3 fatty acids or a placebo.

SECONDARY OUTCOMES:
Hepatic fatty acid partitioning | Eight weeks
  Investigators will measure the contribution of newly synthesised fatty acids and dietary fatty acids to triglyceride production and oxidation pathways in the liver at baseline and 8 weeks after taking n-3 fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Hodson, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Centre for Diabetes, Endocrinology and Metabolism, Oxford, United Kingdom

REFERENCES:
- [Derived] Green CJ, Pramfalk C, Charlton CA, Gunn PJ, Cornfield T, Pavlides M, Karpe F, Hodson L. Hepatic de novo lipogenesis is suppressed and fat oxidation is increased by omega-3 fatty acids at the expense of glucose metabolism. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e000871. doi: 10.1136/bmjdrc-2019-000871. PMID 32188593